CLINICAL TRIAL: NCT07095894
Title: A Randomized Placebo-controlled Trial of Spectacles With Highly Aspherical Lenslets or 0.05% Atropine to Slow Progression of Myopia in Children
Brief Title: A RCT of Spectacles With Aspherical Lenslets or 0.05% Atropine for Myopia Control
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jaeb Center for Health Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MTS2
Record Dates: First submitted 2025-07-21; First posted 2025-07-31 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Myopia
Keywords: myopia; spectacles; atropine; pediatric
MeSH Terms: conditions — Myopia | interventions — Atropine; Eyeglasses

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (4):
- Atropine Group (Experimental): Daily low-concentration atropine (0.05%) eyedrops plus spectacles with single vision lenses (SVL)
  Interventions: Drug: Atropine
- Placebo Group (Placebo Comparator): Daily placebo eyedrops plus spectacles with single-vision lenses (SVL)
  Interventions: Drug: Placebo Eyedrops
- HAL Group (Experimental): Daily placebo eyedrops plus spectacles with highly aspherical lenslets
  Interventions: Device: Spectacles with HAL; Drug: Placebo Eyedrops
- Combined Group (Experimental): Daily low-concentration atropine (0.05%) eyedrops plus spectacles with highly aspherical lenslets
  Interventions: Drug: Atropine; Device: Spectacles with HAL

INTERVENTIONS:
Drug: Atropine — Daily 0.05% atropine eyedrops
  Arms: Atropine Group; Combined Group
Device: Spectacles with HAL — Spectacle lenses with highly aspherical lenslets (HAL)
  Arms: Combined Group; HAL Group
Drug: Placebo Eyedrops — Daily placebo eyedrops
  Arms: HAL Group; Placebo Group

SUMMARY:
To date, randomized trials of low-concentration atropine eyedrops and specially designed spectacle lenses to slow the progression of myopia are limited in number and results are inconsistent in non-Asian children.

Although results of some recent randomized clinical trials outside the US are promising, additional studies in children are needed to test the safety and efficacy of low-concentration atropine and specially designed spectacle lenses as treatments to slow the progression of myopia during the peak years for eye growth.

After a run-in phase to demonstrate adherence with nightly eyedrops (artificial tears) and spectacle correction, children 5 to <12 years old with myopia of 0.75D to 6.00D cycloplegic spherical equivalent refractive error (SER) and at least 0.75D myopia in both principal meridians of each eye will be randomized in a 2x2 factorial design to treatment with 1) nightly 0.05% atropine or placebo eyedrops, and 2) spectacles with highly aspherical lenslets (HAL) or single vision spectacles, and followed every six months for 24 months. Change in axial length over 24 months and change in SER over 24 months are the primary and secondary outcomes, respectively.

All children will return for a visit at 30 months (after 6 months of no treatment other than single-vision spectacles alone between 24 and 30 months).

ELIGIBILITY:
Inclusion Criteria:

1. Age 5 years to <12 years at time of enrollment. Children within 4 weeks of their 12th birthday are not eligible.
2. Refractive error meeting the following by cycloplegic autorefraction:

   * Myopia of 0.75D to 6.00D SER and at least 0.75D in both principal meridians of each eye
   * Astigmatism <2.50D both eyes
   * Anisometropia <1.50D SER
3. Investigator has confirmed the following regarding best-corrected distance visual acuity (VA) in habitual spectacles or trial frames using the investigator's preferred VA testing method:

   * VA is age normal in both eyes1,2
   * 5-6 years: approximately 20/32 or better, ≤ 0.24 logMAR, ≥ 73 letters
   * 7-12 years: approximately 20/25 or better, ≤ 0.14 logMAR, ≥ 78 letters
   * Interocular difference ≤2 logMAR lines (0.2 logMAR) or ≤ 10 letters
4. Wearing spectacles by parent report ≥90% of waking hours ≥30 days duration before enrollment. For children who meet all other inclusion criteria but whose single-vision spectacles are broken or lost within the last 90 days, enrollment can proceed as long as the child was wearing their single-vision spectacles ≥90% of waking hours ≥30 days before the spectacles were broken or lost.
5. Gestational age ≥ 32 weeks.
6. Birth weight >1500 g.
7. Parent(s) and assenting child understand the study procedures and are willing to accept randomization to atropine 0.05%, HAL lenses, atropine combined with HAL lenses, or placebo (i.e., neither active treatment).
8. Parent is willing to participate in a 2- to 4-week run-in phase using nightly artificial tear eyedrops in both eyes.
9. Family can return in 2 to 4 weeks for possible randomization.
10. Child is willing to refrain from contact lenses for the duration of the study.
11. Parent has a phone (or access to a phone) and is willing to be contacted by the clinical site staff.
12. Relocation outside of the area of an active PEDIG site within the next 32 months is not anticipated.

Exclusion Criteria:

1. Current or previous pharmacologic or light therapy used for myopia treatment.
2. Current or prior contact lens wear more than 7 days in the past 12 months
3. Current or previous use of bifocals, progressive-addition lenses, multi-focal contact lenses, or focus- or contrast-modifying spectacle lenses.
4. Current or previous use of orthokeratology, rigid gas permeable, or other contact lenses used to slow myopia progression.
5. Current or previous myopia control treatment or other uses of atropine, pirenzepine or other anti-muscarinic agents.
6. Known atropine allergy
7. Abnormality of the cornea, lens, central retina, iris, or ciliary body
8. Current constant or intermittent strabismus (phorias are acceptable)
9. Verified history of amblyopia or nystagmus.
10. Prior strabismus, intraocular, or refractive surgery
11. Down syndrome or cerebral palsy
12. Diseases known to affect accommodation, vergence, or ocular motility (e.g., multiple sclerosis, Graves' disease, myasthenia gravis, diabetes mellitus)
13. Any condition that, in the judgment of the investigator, could influence refractive error development.
14. Existing conditions in the opinion of the investigator that may affect the long-term health of the eye or require regular pharmacologic treatment that may adversely interact with study medication (e.g., JIA, glaucoma, pre-diabetes).
15. Inability to comprehend and/or perform any study-related procedures.
16. Individuals who are pregnant, lactating, or intending to become pregnant within the next 30 months.

    a. A negative urine pregnancy test at randomization and the 6-, 12-, 18-, and 24-month follow-up visits will be required for individuals who have experienced menarche (at least one menstrual cycle).
17. Immediate family member (spouse, biological or legal guardian, child, sibling, parent) who is investigative site personnel directly affiliated with this study or who is an employee of the Jaeb Center for Health Research.
18. Sibling of, or living in the same household as, another child who is concurrently enrolled in the study.
19. Allergy to benzalkonium chloride (eyedrop preservative).

Ages: 5 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 348 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2028-12-01 (Estimated); Study Completion 2029-06-01 (Estimated)

PRIMARY OUTCOMES:
Primary efficacy outcome - change in axial length | 24 months.
  Change in axial length from baseline to 24 months (on-treatment) as measured by a masked examiner using cycloplegic biometry.

CONTACTS AND LOCATIONS:
Overall Officials: Lori Ann F Kehler, OD, Study Chair — Vanderbilt University Medical Center; Katherine A Lee, MD, PhD, Study Chair — Jaeb Center for Health Research

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF

DOCUMENTS (3):
  • Study Protocol (2025-06-12): https://cdn.clinicaltrials.gov/large-docs/94/NCT07095894/Prot_000.pdf
  • Statistical Analysis Plan (2025-07-15): https://cdn.clinicaltrials.gov/large-docs/94/NCT07095894/SAP_001.pdf
  • Informed Consent Form (2025-06-30): https://cdn.clinicaltrials.gov/large-docs/94/NCT07095894/ICF_002.pdf